CLINICAL TRIAL: NCT01198743
Title: Search for the Presence of Genetic Alteration in the Plasma of Patients With Stage II-III Colorectal Cancers: Prognosis Impact
Brief Title: Presence of Circulating Tumor DNA in Colorectal Cancer
Acronym: ALGECOLS
Status: Completed | Type: Observational
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Other Study IDs: P040433
Record Dates: First submitted 2010-06-02; First posted 2010-09-10 (Estimated); Last update posted 2017-08-29 (Actual); Status verified 2017-08

CONDITIONS: Colorectal Neoplasms
Keywords: Genetics modifications; colorectal cancer; prognosis aim; DNA; Plasma
MeSH Terms: conditions — Colorectal Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — serum and tissue
Oversight: Data Monitoring Committee: No

SUMMARY:
Cancer is a DNA disease characterized by the presence of genetics alterations in cancer cells.

The recent studies underline that these recurring alterations must be considered as a good molecular marker. In fact, they could use for tumor DNA detection in different biological fluids.

So, the main purpose is to define the presence of circulating tumor DNA in the patients plasma with colorectal cancer, by the presence of mutation (KRAS, NRAS, BRAF, APC, TP53 and MIRCOSATELLIE instability).

These molecular analysis will be done both in tumor and plasma samples,

This trial allows to characterize the prognostic value of circulating tumoral DNA presence in colorectal cancer.

DETAILED DESCRIPTION:
Two major issues appear in improving the prognosis of cancer patients, the first is early detection and the second is the risk of recurrence or the early diagnosis of recurrence in order to propose the most appropriate treatment for patients.

Cancer is a DNA disease that is characterized by the acquisition by the tumor cell during carcinogenesis of a number of recurrent genetic alterations. The development of molecular tools that can easily characterize these abnormalities specific to tumor cells, allows us to consider their use in clinical practice. These genetic alterations could represent useful molecular markers for detecting the presence of tumor DNA in various biological fluids including plasma of cancer patients. This circulating tumor DNA, whose nature is confirmed by the similarity of genetic alterations with those observed from DNA extracted from tumor cells of the patients, represents a molecular marker of cancer available from a single sample and could be an alternative to the use of more conventional markers such as CEA. We propose in this study to confirm the predictive value on the risk of recurrence or metastasis of circulating tumor DNA in plasma of patients with colorectal cancer from a cohort study (250 patients with non-metastatic colorectal cancer (Stage II and III). This is a multicenter prospective study. The cohort of patients will be followed for a minimum period of 36 months. A biological analysis of the tumor in search for the main genetic alterations of colorectal cancer cells will be made (KRAS, NRAS, TP53, BRAF and APC mutations as well as the presence of a microsatellite instability). These same genetic alterations will be sought on a plasma sample taken before surgery and during follow-up (9 samples in total). The objectives of this study will be 1/to assess the prognostic value of the presence of circulating tumor DNA in plasma, by searching for an association between the risk of and the presence of genetic alteration in the plasma of these patients, 2/to search for a relationship between initial rate of circulating tumor DNA and the risk of local recurrence,3/ to characterize the relationship between the type of alterations in the plasma at the initial diagnosis of circulating tumor DNA and the risk of recurrence 4/ to assess during the follow-up the prognostic value of the occurrence of tumor circulating DNA.

ELIGIBILITY:
Inclusion Criteria:

* patients aged Superior to 18 and inferior to 85
* Colon or rectal cancer stage II and III should be surgically treated
* informed consent signed

Exclusion Criteria:

* patients suffered from synchronous metastasis disease in initial cancer diagnosis
* patients with 2 synchronous colorectal cancers
* receiving chemotherapy or radiotherapy, before operation

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: defined population : patients suffer from colorectal cancers in stage II-III
Sampling Method: Non-Probability Sample
Enrollment: 261 (Actual)
Dates: Start 2005-11; Primary Completion 2017-05 (Actual); Study Completion 2017-05 (Actual)

PRIMARY OUTCOMES:
local recidivism or metastasis reappearance | 6 months after operation

SECONDARY OUTCOMES:
specificity and global safety | 36 monhs after operation

CONTACTS AND LOCATIONS:
Overall Officials: Pierre LAURENT-PUIG, Principal Investigator — HEGP/ Paris Descartes University
Locations (1):
- HEGP, Paris, France